CLINICAL TRIAL: NCT05228665
Title: HEART Rate Variability Biofeedback in LOng COVID-19 (HEARTLOC)
Acronym: HEARTLOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: University of Manchester (Other); Leeds Comunity Healthcare NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Manoj Sivan, Associate Professor and Consultant in Rehabilitation Medicine, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 304567
Record Dates: First submitted 2022-01-30; First posted 2022-02-08 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: Long Covid; Post-Covid Syndrome; Post-Covid Condition; Post-Acute Covid Syndrome; Autonomic Nervous System
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective cohort (Experimental): Participants will be shown a paced breathing programme and instructed to implement this for 10 minutes twice daily for 4 weeks. During the 10-minute breathing exercises, the participant will need to wear the Polar H10 chest strap and can remove this when finished. The breathing will ideally be a breathing pattern of a 4-second nasal inhale, and 6-second nasal exhale using the 'resonance' programme in the 'biofeedback' section of EliteHRV app. They will be advised to monitor the graph of HRV on EliteHRV which allows real-time assessment of HRV and to aim to breathe in and out deeply to raise the HRV graph reading as much as possible each time. They will be advised to perform the breathing programme lying down with minimal distractions on waking in the morning and just before bed in the evening, preferably in the same location each time.
  Interventions: Behavioral: Heart Rate Variability Biofeedback (HRV-B)

INTERVENTIONS:
Behavioral: Heart Rate Variability Biofeedback (HRV-B) — Breathing technique twice every day (10 min each) to increase HRV

SUMMARY:
Long COVID is a common but highly debilitating illness which develops after infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2 or COVID-19). It is thought to affect as many as 1 in 7 people following COVID-19 infection. It can produce a vast array of symptoms including fatigue, breathlessness, fast heart rate, blood pressure disturbance, temperature disturbance, and dry mouth. Many of these symptoms could be explained by the nervous system being predominantly in a stress or 'fight or flight' response, also known as dysautonomia. One way of assessing whether this is the case is by measuring heart rate variability (HRV). This is the time variation between heart beats and is a marker of how stressed the nervous system is or how strong is the 'fight or flight' response. Heart rate variability can be measured using devices which are worn round the wrist or attach to the chest. An increased variability in heart rate corresponds with a more relaxed nervous system and decreased variability with a more stressed nervous system. Monitoring HRV in real-time and implementing interventions such as a breathing regime to maximise HRV is known as HRV biofeedback. The body can be trained out of the fight or flight response and into the 'rest and digest' mode response of the nervous system in this way and potentially significantly improve symptoms. We propose that for people with Long COVID, a programme of structured breathing exercises over 4 weeks whilst tracking HRV can demonstrate an improvement in HRV and consequently improve Long COVID symptoms.

DETAILED DESCRIPTION:
Participants will be shown a paced breathing programme and instructed to implement this for 10 minutes twice daily for 4 weeks. During the 10 minute breathing exercises, the participant will need to wear the Polar H10 chest strap and can remove this when finished. The breathing will ideally be a breathing pattern of a 4 second nasal inhale, and 6 second nasal exhale using the 'resonance' programme in the 'biofeedback' section of EliteHRV app. Researchers will monitor the participant's comfort and ease during this breathing demonstration, if participants find this breathing rate too slow then it can be tailored to ensure a tolerable slow breathing rate with minimal impact on symptoms - most likely by reducing both inhale and exhale in 1 second increments until a more tolerable breathing rate and pattern is found. They will be advised to monitor the graph of HRV on EliteHRV which allows real-time assessment of HRV and to aim to breathe in and out deeply to raise the HRV graph reading as much as possible each time. Participant Information Sheet provides more clarification and instruction on this. They will be advised to perform the breathing programme lying down with minimal distractions on waking in the morning and just before bed in the evening, preferably in the same location each time. During this 4 week period researchers will make weekly contact by phone to check progress and help resolve any queries. The participant will also have contact details of the researchers in case of any technical issues with Polar H10 chest strap or app during the 4 week study period.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Confirmed Long COVID based on a positive PCR or antibody test and Long COVID symptoms as per the NICE criteria for post-COVID syndrome
* Current Leeds COVID Rehabilitation service user
* Self-rating of 'moderate/severe' on the Leeds COVID Rehabilitation Service Long COVID participant reported outcome measure (known as C19-YRS)
* Abnormal NASA Lean Test (NLT)

Exclusion Criteria:

* Age < 18 years
* Unable to use the wearable or smartphone app technology
* Cognitive problems or mental health disorders causing inability to consent
* Cardiac arrhythmia (current or prior tachyarrhythmia or bradyarrhythmia)
* Existing significant cardiorespiratory disease which might be expected to affect studied symptoms of palpitations, presyncope, breathlessness and fatigue (asthma not included in this definition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Modified C19-YRS (COVID-19 Yorkshire Rehabilitation Scale) | Up to 6 weeks
  The C19-YRSm will be completed by the patient every week for a total of 6 weeks. There will be a total of 7 C19-YRSm documents completed. The C19-YRSm consists of 17 items with each item rated on a 4-point numerical rating scale from 0 (no symptom) to 3 (life disturbing or affecting all aspects of daily life). The C19-YRSm is divided into four subscales (range of total score for each subscale): symptom severity score (0-30), functional disability score (0-15), other symptoms (0-25), and overall health (0-10). A higher score for the first 3 subscores represents higher severity. Conversely, a lower overall health score represents greater severity.

SECONDARY OUTCOMES:
HRV (Heart Rate Variability) score | Up to 6 weeks
  We will be collecting both medium and short term HRV data. Participants will wear a Fitbit for 6 weeks which will collect HRV data whilst sleeping each night, thus collecting 6 weeks of consecutive nocturnal HRV data. In addition they will wear a Polar H10 chest strap for 10 minutes twice daily whilst performing breathing exercises to collect frequent short-term HRV data. For both data sets an increase in HRV is expected as this denotes an improvement in heart rate variability.
  Fitbit measures HRV in milliseconds on a scale from 0 to 100 (or more if HRV exceeds 100ms) A higher score represents more variability and therefore improvement.
  The Elite HRV also provides a score of HRV on a scale from 0 to 100 with a higher score representing improvement. The score is derived from the root mean square of successive differences between heartbeats in milliseconds (rMSSD).

OTHER OUTCOMES:
COMPASS 31(Composite Autonomic Symptom Score) | Up to 6 weeks
  The COMPASS 31 will be completed by the participant at the initial visit and again 6 weeks later at the end of the study. Autonomic symptoms are scored for different domains including orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder and pupillomotor. Total scores for each domain are multiplied by a set weighting and then added together to provide a score out of 100 representing severity of autonomic symptoms. A higher score represents greater severity
EQ5D-5L(EuroQol Five Dimension Quality of Life) | Up to 6 weeks
  The EQ5D-5L will be completed by the participant at the initial visit and again 6 weeks later at the end of the study. 4 domains are assessed on a scale of 1 to 5: mobility, self-care, usual activities, pain/discomfort and anxiety and depression. A greater score represents greater severity. In addition participants self-rate their overall health on a scale f 0 to 100. 100 represents best health possible and 0 represents worst health possible.
aAP(Adapted Autonomic Profile) | Up to 6 weeks
  Participant will complete an aAP at initial visit and again 6 weeks later at the end of the study. This test has binary outcome: normal or abnormal. There is no score generated by the test. We will assess whether those deemed normal or abnormal at the beginning change as a result of the intervention.
World Health Organisation Disability Assessment Schedule (WHODAS) | Up to 6 weeks
  This is validated generic measure of functioning and disability. The 36-item scale captures six domains of life (cognition, mobility, self-care, getting along, life activities and participation) with a summary score ranging from 0 (no disability) to 100 (full disability)

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Sivan, MD, Principal Investigator — University of Leeds
Locations (1):
- Leeds Community Healthcare NHS Trust, Leeds, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available on requesting the corresponding author
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After completion of data collection from 30 participants
Access Criteria: Open Science Framework registration
URL: https://osf.io/

REFERENCES:
- [Derived] Corrado J, Iftekhar N, Halpin S, Li M, Tarrant R, Grimaldi J, Simms A, O'Connor RJ, Casson A, Sivan M. HEART Rate Variability Biofeedback for LOng COVID Dysautonomia (HEARTLOC): Results of a Feasibility Study. Adv Rehabil Sci Pract. 2024 Jan 28;13:27536351241227261. doi: 10.1177/27536351241227261. eCollection 2024 Jan-Dec. PMID 38298551
- [Derived] Corrado J, Halpin S, Preston N, Whiteside D, Tarrant R, Davison J, Simms AD, O'Connor RJ, Casson A, Sivan M. HEART rate variability biofeedback for long COVID symptoms (HEARTLOC): protocol for a feasibility study. BMJ Open. 2022 Nov 21;12(11):e066044. doi: 10.1136/bmjopen-2022-066044. PMID 36410797